CLINICAL TRIAL: NCT04686747
Title: COVID - 19 and Advanced Gastro-intestinal Cancer Treatment
Acronym: COVID - AGICT
Status: Completed | Type: Observational
Sponsor: S.M. Misericordia Hospital (Other)
Responsible Party: Principal Investigator, Giuliani Giuseppe, MD, Ospedale della Misericordia
Other Study IDs: MH - COVID - AGICT
Record Dates: First submitted 2020-12-26; First posted 2020-12-29 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cancer; Gastric Cancer; Esophagus Cancer; Colorectal Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Esophageal Cancer
- Gastric Cancer
- Pancreatic Cancer
- Colorectal Cancer

SUMMARY:
A multicenter Italian retrospective study on COVID-19 pandemic condition and advanced Gastro - Intestinal Cancer.

Are in Italy increased the new diagnosis of GI cancer in advanced stage in the 2020 compared with 2019, as a consequence of COVID-19?

DETAILED DESCRIPTION:
1. Background The ongoing COVID-19 pandemic condition had a catastrophic consequence on the healthcare system. In order to contain the death from other diseases, such as cancer, the healthcare system still fights a challenging battle focusing the attention on COVD-19 without losing sight of other patient care. Routine screening and non urgent surgeries reduced to increase capacity for COVID-19 patients complications. Moreover, it must take into account the fear for COVID-19 exposure of patients during the routine assessments.

   Nevertheless, death related to other causes is not decreased. Standard cancer screening is decreased, such as colorectal cancer protocol which dropped by 84.5% through May 20201. As a consequence, according to London JW et al, the incidence of new cancer diagnoses decreased of 65.2%. As matter of fact, the new diagnosis of melanoma dropped by 67.1%, as well as the new diagnosis of lung cancer which dropped of 46.8%1 in April 2020 compared to one year earlier. Furthermore, the number of advanced gastrointestinal cancers are supposed to be increased in the surgical community. As conventional wisdom, the number of patients with locally advanced or metastatic gastrointestinal, as well as patients needing an emergency or a palliative procedure (i.e., stoma, feeding jejunostomy, gastroentero anastomosis) seems increased this year compared to 2019. These therapeutic delays may influence the long-term survival of these patients. An increased rate of related death is expected, rising from 15.5% to 16.6% and 4.8% to 5.3 % for colorectal and lung cancer, respectively. This study aims to investigate whether the main gastrointestinal cancers was diagnosed in a more advanced stage in 2020 compared to 2019 as a consequence of Covid-19 pandemic.
2. Methods This is a multicenter retrospective study that will include patients treated for esophageal, gastric, pancreatic and colorectal cancer, from January 2019 to December 2020 in more than 50 Italian centers. All patients will be included in a disease-specific database, which will be sent to each Italian reference center. A minimum of 1.000 patient/year is expected to show a significative difference between the considered years.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to elective surgery for esophageal, gastric, pancreatic and colorectal cancer in the year 2019-2020;
* Patients submitted to emergency surgery/procedure (Interventional radiology, endoscopic procedure) for complication (i.e. perforation, bleeding, occlusion) secondary to esophageal, gastric, pancreatic and colorectal cancer in the year 2019-2020;
* Patients submitted to palliative surgery/procedure (i.e. stoma, GEA, external biliary drainage, feeding jejunostomy) for esophageal, gastric, pancreatic and colorectal cancer in the year 2019-2020;
* Patients undergoing preoperative chemo or radiation therapy for locally advanced or metastatic esophageal, gastric, pancreatic and colorectal cancer in the year 2019-2020;
* Patients undergoing to adjuvant therapy after esophageal, gastric, pancreatic and colorectal cancer I surgery in the year 2019-2020

Exclusion Criteria:

* Patients under 18 years old and over 85 years old;
* Patients with multiple tumors.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a multicenter retrospective study that will include patients treated for esophageal, gastric, pancreatic and colorectal cancer, from January 2019 to December 2020 in more than 50 Italian centers. In the study are included both patients treated with a curative or palliative intent.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of advanced Esophageal, Gastric, Pancreatic and Colorectal cancer in 2020 compared to 2019. | From January 2019 to December 2020
  The primary endpoint is to show if in Italy the number of cancer mentioned above, was diagnosed in a more advanced stage (i.e. > I stage, Metastatic disease) in 2020 compared to 2019 as a consequence of COVID-19 pandemic condition.

SECONDARY OUTCOMES:
Rate of neo-adjuvant therapy in 2020 compared to 2019 | From January 2019 to December 2020
  To show any difference in the rate of cancer related neo-adjuvant therapy in 2020 compared to 2019;
Rate of palliative procedure in 2020 compared to 2019 | From January 2019 to December 2020
  To show any difference in the rate of cancer related palliative procedures/ bridge therapy in 2020 compared to 2019, before starting with standard treatment;
Rate of preoperative chemo or radiotherapy in 2020 compared to 2019 for metastatic disease. | From January 2019 to December 2020
  To show any difference of patients unable to performer cancer related preoperative chemo or radiotherapy in 2020 compared to 2019 due to scarce performance status or for symptomatic disease;
Rate of patient unable to performer adjuvant treatment in 2020 compared to 2019 | From January 2019 to December 2020
  Rate of patients unable to performer cancer related adjuvant therapy in 2020 compared to 2019 due to scarce performance status

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General and Emergency Surgery. Misericordia Hospital. Director: Coratti Andrea, MD, Grosseto, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giuliani G, Coletta D, Guerra F, Esposito S, Esposito A, De Pastena M, Rega D, Delrio P, La Raja C, Spinelli A, Massaron S, De Nardi P, Kauffmann EF, Boggi U, Deidda S, Zorcolo L, Marano A, Borghi F, Piccoli M, Depalma N, D'Ugo S, Spampinato M, Cozzani F, Del Rio P, Marcellinaro R, Carlini M, De Rosa R, Scabini S, Maiello F, Polastri R, Turri G, Pedrazzani C, Zese M, Parini D, Coratti A; MIS-COVID-AGICT Collaborative Group. The MIS-COVID-AGICT Study: Trend of Minimally Invasive Surgery for Gastrointestinal Cancer Treatment During the First Waves of the COVID-19 Pandemic in Italy. Subgroup Analysis from the COVID-AGICT Study: COVID-19 and Advanced Gastrointestinal Cancer Surgical Treatment. J Laparoendosc Adv Surg Tech A. 2023 Jun;33(6):579-585. doi: 10.1089/lap.2023.0058. Epub 2023 May 2. PMID 37130329